CLINICAL TRIAL: NCT00131508
Title: A Randomized Controlled Trial of Oral Glutamine Supplementation Versus a Placebo Supplement in Children With Sickle Cell Anemia
Brief Title: Trial of Oral Glutamine in Patients With Sickle Cell Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow participant accrual
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCGLU2
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2010-03

CONDITIONS: Anemia, Sickle Cell
Keywords: Hemoglobin S Disease; Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): Glutamine
  Interventions: Drug: Glutamine
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glutamine — 0.6 gm/kg of oral glutamine per day, in two doses for one year.
  Arms: 2
Drug: Placebo — Placebo
  Arms: 1

SUMMARY:
Children with sickle cell anemia (SCA) seem to have higher energy needs than children who do not have the disease. This may be the reason why children and teenagers with sickle cell anemia tend to be smaller, weigh less, and have less fat and muscle than children and teens that do not have the disease.

This study is being done to find out if giving a supplement called glutamine will help children with sickle cell anemia by lowering their energy needs and improving their growth and strength. Children will be randomly assigned (like a flip of a coin) to one of two groups. One group will take glutamine and one group will take a placebo (a protein mixture that looks like glutamine but may not have the same effect in the body). No one will know which group is taking which supplement until the study has been completed. Children will be in the study for 12 months.

DETAILED DESCRIPTION:
1. The study will compare the effect of glutamine and placebo on resting energy expenditure (REE) in children with sickle cell anemia (SCA) by comparing the change in REE ratio between baseline and 12 months.
2. The study investigates the effect of oral glutamine and placebo on body composition in children with SCA by comparing the difference in body mass indexes (BMIs) and percent of body fat (DEXA Scan) between baseline and 12 months of treatment in the two groups.
3. This Study will investigate the effect of oral glutamine and placebo on growth in children with SCA by comparing the Z scores for one year before baseline to 1 year while on study.
4. This study will investigate the effect of oral glutamine and placebo in children with SCA by comparing the difference in the levels of plasma and red blood cell glutamine between baseline and 12 months of treatment in the two groups.
5. This study will investigate the clinical effects (strength and exercise endurance) of oral glutamine and placebo in children with SCA by comparing the difference between baseline and 12 months of treatment in the two groups.
6. This study will evaluate quality of life in children with SCA who have glutamine or placebo for 12 months.
7. This study will evaluate the changes in REE over time in a small group of patients that will have REE measurement at months 3, 6, and 9. This objective will be offered to all patients, but will be "additional studies" that are not required to participate in the protocol.

ELIGIBILITY:
Inclusion Criteria:

Active patient (presently receiving medical care for SCA) at the St. Jude Comprehensive Sickle Cell Center (SJCSCC) or an affiliate or alliance of St Jude. Patient must not be in the high risk category as defined by the SJCSCC. High risk is defined as follows:

* 3 or more admissions and/or emergency department visits for pain within the past 12 months, or;
* 2 or more episodes of acute chest syndrome within the past 24 months, or;
* A combination of pain and ACS events > 3 within the past 12 months.
* 5-18 years of age
* Diagnosis of Hb SS or HB0Thal
* Weight >15 kg
* <50th percentile for height/age or weight/age or weight/ height, or <90% ideal body weight, or <90% of BMI for age/ gender.
* Is willing to sign informed consent

Exclusion Criteria

* Patients receiving hydroxyurea or any other anti-sickling agent, chronic transfusion, or nutrition supplements.A nutrition supplement is any high calorie or high protein food additive or oral supplement being used for the purpose of weight gain.
* History of poor compliance (Missing two or more clinic appointments in the past year).
* Renal or liver dysfunction
* Renal dysfunction as defined by serum creatinine >1.5 times normal for age based on testing lab.
* Hepatic dysfunction as defined by alanine aminotransferase (ALT) >2 times the upper limit of normal for age based on testing lab.
* Breastfeeding
* Pregnancy.Females of childbearing potential must have negative serum or urine pregnancy test (record date of test).
* Patients enrolled on previous glutamine protocol (SCDGLU).
* Patients who are considered high risk

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2004-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Williams, MS, RD, EdD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 participants were recruited from July, 2004 through October, 2007.
Pre-assignment Details: 25 of the 27 participants were randomized to either the Glutamine or Placebo arm.
Groups:
- Placebo: A mixture of non-essential amino acids containing glycine, alanine, and serine.
- Glutamine: Glutamine dosage of 0.60 gm/kg body weight per day divided into two doses.
Period: Overall Study
Arm/Group | Placebo | Glutamine
Started | 12 | 13
Completed | 9 | 5
Not Completed | 3 | 8
Not completed — Disease progression | 0 | 2
Not completed — Non-Compliance | 2 | 4
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Glutamine | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (2.9) | 9.1 (3.6) | 9.1 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting Energy Expenditure From Baseline to 12 Months
Description: To compare the effect of glutamine and placebo on resting energy expenditure (REE) in children with sickle cell anemia (SCA) by comparing the change in REE ratio between baseline and 12 months. REE was measured by indirect calorimetry, using a metabolic cart.REE Ratio =(REE Measured/REE Predicted)x 100).Change was defined as 12 Month REE Ratio minus Baseline REE Ratio.The REE Ratio was evaluated at baseline and 12 months.The REE Ratio is calculated as (REE Measured / REE Predicted) x 100).REE units are measured as (Kcal / day).Change was defined as 12 Month REE Ratio minus Baseline REE Ratio.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: REE ratio
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 12 | 13
REE ratio | -5.5 [-37.6 to 12.2] | 7.1 [-9.0 to 41.3]
Statistical Analysis 1: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change in REE ratio between the placebo and glutamine groups. The study was designed to provide 80% power at an alpha level of 0.05 for this objective. Due to slow accrual, the sample size of 46 participants required to obtain the designed power of the study was not realized; Test type: Superiority or Other; p = 0.17, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Body Mass Index From Baseline to 12 Months
Description: To investigate the effect of oral glutamine and placebo on body composition in children with SCA by comparing the difference in body mass indexes (BMI) between baseline and 12 months of treatment in the two groups.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: kg/m2
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 12 | 13
kg/m2 | 0.1 [-0.3 to 1.2] | 0.8 [-0.6 to 0.9]
Statistical Analysis 1: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change of body mass index between the placebo and glutamine groups; Test type: Superiority or Other; p = 0.53, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Red Blood Cell Glutamine From Baseline to 12 Months
Description: To investigate the effect of oral glutamine and placebo in children with Sickle Cell Anemia (SCA) by comparing the difference in the levels of red blood cell glutamine between baseline and 12 months of treatment in the two groups.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: nmol/mg creatinine
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 12 | 13
nmol/mg creatinine | 43.5 [-173.9 to 137.0] | 100.8 [21.1 to 262.4]
Statistical Analysis 1: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change in red blood cell glutamine between the placebo and glutamine groups; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Quality of Life Measures From Baseline to 12 Months.Scores for Each Subcategory Range From 0 (Best) to 4 (Worst).This is True for Both Patient and Parent Reports.
Description: Evaluation of quality of life at baseline and 12 months in the glutamine versus placebo group using the PedsQL Version 4.0 inventory. This instrument measures individual well being across physical, emotional, social, and school function categories using patient self-reports and/or parent reports. The tool contains a 15-question, age-specific, self-report inventory (for children age 5-7 years, 8-12 years, and 13-18 years) and a corresponding parent inventory. Lower scores indicate a better quality of life.
Time Frame: Baseline and 12 Months
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 12 | 13
Units on a scale
  Baseline Parent Reported Physical Function | 1.4 [0.3 to 3.5] | 2.0 [0.0 to 2.9]
  Baseline Parent Reported Emotional Function | 1.0 [0.0 to 2.0] | 2.0 [0.0 to 4.0]
  Baseline Parent Reported Social Function | 0.6 [0.0 to 2.6] | 1.8 [0.0 to 3.0]
  Baseline Parent Reported School Function | 1.8 [0.8 to 2.6] | 2.0 [0.0 to 3.6]
  12 Months Parent Reported Physical Function | 2.5 [0.3 to 3.3] | 2.1 [0.5 to 2.9]
  12 Months Parent Reported Emotional Function | 1.4 [0.0 to 2.0] | 1.2 [0.0 to 2.2]
  12 Months Parent Reported Social Function | 2.0 [0.0 to 2.8] | 1.2 [0.4 to 2.4]
  12 Months Parent Reported School Function | 1.8 [0.4 to 3.2] | 2.4 [1.6 to 3.8]
  Baseline Participant Reported Physical Function | 0.9 [0.4 to 2.8] | 1.0 [0.1 to 2.0]
  Baseline Participant Reported Emotional Function | 0.8 [0.0 to 2.6] | 1.2 [0.0 to 2.0]
  Baseline Participant Reported Social Function | 1.0 [0.0 to 2.0] | 1.2 [0.0 to 2.8]
  Baseline Participant Reported School Function | 1.6 [0.8 to 2.8] | 1.3 [0.0 to 2.4]
  12 Months Participant Reported Physical Function | 1.0 [0.5 to 2.1] | 1.0 [0.6 to 2.9]
  12 Months Participant Reported Emotional Function | 0.8 [0.0 to 2.0] | 1.2 [0.0 to 3.6]
  12 Months Participant Reported Social Function | 1.2 [0.4 to 2.2] | 1.0 [0.0 to 3.6]
  12 Months Participant Reported School Function | 1.6 [1.0 to 3.2] | 1.8 [1.0 to 3.4]
Statistical Analysis 1: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between baseline parent reported physical function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between baseline parent reported emotional function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between baseline parent reported social function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between baseline parent reported school function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between 12 month parent reported physical function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between 12 month parent reported emotional function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.65, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between 12 month parent reported social function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between 12 month parent reported school function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between baseline patient reported physical function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between baseline patient reported emotional function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.99, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between baseline patient reported social function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between baseline patient reported school function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between 12 month patient reported physical function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between 12 month patient reported emotional function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between 12 month patient reported social function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change between 12 month patient reported school function in the placebo and glutamine groups; Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Height Z-score From Baseline to 12 Months
Description: To investigate the effect of oral glutamine and placebo on height Z-score in children with Sickle Cell Anemia (SCA) between baseline and 12 months on treatment.
Time Frame: Baseline and 12 months
Population: Analyzed patients had a height measurement at both baseline and 12 months.
Measure: Median (Full Range); unit: Z-score
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 9 | 5
Z-score | -0.1 [-52.2 to 0.4] | 0.0 [-0.2 to 0.3]
Statistical Analysis 1: Comparison: Placebo; We tested the null hypothesis that the median difference in height Z-Score betweeen baseline and 12 months is equal to zero versus the alternative hypothesis that the difference is not zero; Test type: Superiority or Other; p = 0.20, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Glutamine; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.81, Wilcoxon Signed Rank Test
Statistical Analysis 3: Comparison: Placebo vs Glutamine; We tested the null hypothesis that the median difference in height Z-Score betweeen baseline and 12 months differs between the Glutamine and Placebo groups; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Height Percentile From Baseline to 12 Months
Description: To investigate the effect of oral glutamine and placebo on height percentile in children with Sickle Cell Anemia (SCA) between baseline and 12 months on treatment.
Time Frame: Baseline and 12 months
Population: Analyzed patients had a height measurement at both baseline and 12 months.
Measure: Median (Full Range); unit: Percentile
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 9 | 5
Percentile | 0.0 [-12.5 to 20.0] | 0.0 [-12.5 to 14.5]
Statistical Analysis 1: Comparison: Placebo; We tested the null hypothesis that the median difference in height percentile between baseline and 12 months is equal to zero versus the alternative hypothesis that the difference is not zero; Test type: Superiority or Other; p = 0.69, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Glutamine; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.75, Wilcoxon Signed Rank Test
Statistical Analysis 3: Comparison: Placebo vs Glutamine; We test the null hypothesis that the median difference in height percentile between baseline and 12 months differs between the Glutamine and Placebo groups; Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Weight Percentile From Baseline to 12 Months
Description: To investigate the effect of oral glutamine and placebo on weight in children with Sickle Cell Anemia (SCA) between baseline and 12 months on treatment.
Time Frame: Basline and 12 months
Population: Analyzed patients had a height measurement at both baseline and 12 months.
Measure: Median (Full Range); unit: Percentile
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 9 | 5
Percentile | 0.0 [-11.0 to 12.5] | 7.5 [-12.5 to 12.5]
Statistical Analysis 1: Comparison: Placebo; We tested the null hypothesis that the median difference in weight percentile between baseline and 12 months is equal to zero versus the alternative hypothesis that the difference is not zero; Test type: Superiority or Other; p = 0.56, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Glutamine; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 1.0, Wilcoxon Signed Rank Test
Statistical Analysis 3: Comparison: Placebo vs Glutamine; We test the null hypothesis that the median difference in weight percentile between baseline and 12 months differs between the Glutamine and Placebo groups; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Pulse Rate From Baseline to 12 Months
Description: To investigate the clinical effects of oral glutamine and placebo on pulse rate in children with Sickle Cell Anemia (SCA) by comparing the difference between baseline and 12 months of treatment between the two groups.
Time Frame: Baseline and 12 months
Population: Analyzed patients had a height measurement at both baseline and 12 months.
Measure: Median (Full Range); unit: Beats per minute (BPM)
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 7 | 3
Beats per minute (BPM) | 11 [-22 to 44] | 17 [-16 to 34]
Statistical Analysis 1: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change in pulse rate between the placebo and glutamine groups; Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Hand Grip From Baseline to 12 Months.
Description: To investigate the clinical effects of oral glutamine and placebo on hand grip in children with Sickle Cell Anemia (SCA) by comparing the difference between baseline and 12 months of treatment between the two groups.
  Hand grip strength is a measure of muscle strength.Units are measured in Kg.Muscle strength is measured using a hydraulic hand-held dynamometer.Change was defined as 12 Month measure minus baseline.Muscle strength is measured using the hand grip strength via a hydraulic hand-held dynamometer (Kg).
Time Frame: Baseline and 12 months
Population: Analyzed patients had a height measurement at both baseline and 12 months.
Measure: Median (Full Range); unit: kg
Arm/Group | Placebo | Glutamine
Number analyzed (Participants) | 6 | 3
kg | 12 [-3 to 19] | 5 [3 to 12]
Statistical Analysis 1: Comparison: Placebo vs Glutamine; We tested for a significant difference in the median change in hand grip between the placebo and glutamine groups; Test type: Superiority or Other; p = 0.40, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline through 12 months for an average of one year.
Description: Patients were monitored for adverse events throughout the entire course of the study from baseline through 12 months for an average of one year.
Arm/Group | Placebo | Glutamine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

LIMITATIONS AND CAVEATS:
The study was designed to enroll 46 participants (23 per arm). Due to slow accrual the study was terminated after enrolling 27 participants. Of the 27 participants enrolled, 2 dropped out of the study prior to randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes